CLINICAL TRIAL: NCT03386292
Title: Prevalence and Risk Factors for Urinary and Anal Incontinence in Tunisian Middle Aged Women
Brief Title: Urinary and Anal Incontinence in Tunisian Women
Status: Completed | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Syrine GALLAS, Principal investigator, University of Monastir
Other Study IDs: Monastir University
Record Dates: First submitted 2017-12-16; First posted 2017-12-29 (Actual); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Woman
Keywords: prevalence; urinary incontinence; anal incontinence; risk factors; women
MeSH Terms: conditions — Urinary Incontinence; Encopresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
The publications on prevalence and risk factors of urinary and anal incontinence in women were performed mainly in Europe and America. Consequently, result extrapolation to Tunisian population may not be a good practice which justifies this study and demonstrates its importance.

DETAILED DESCRIPTION:
A cross-sectional study will be conducted among female doctors and nurses randomly selected from 3 large hospitals in the center of Tunisia. The prevalence of urinary incontinence and anal incontinence will be measured using validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Professional seniority in the current service over than 6 months
* Subject has given his consent

Exclusion Criteria:

* Resident
* Intern
* An ongoing pregnancy
* A recent birth (less than 6 months)
* A psychiatric disease
* An acute or chronic kidney disease
* Neurological disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female doctors and nurses working at Sahloul Hospital, Taher Sfar Hospital and Fattouma Bourguiba Hospital
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of urinary incontinence | 1 month
  The participant will be asked to fill out the urinary symptom profile questionnaire (USP). This questionnaire contains 13 items to assess stress urinary incontinence, urge urinary incontinence and dysuria. Each question is scored from 0 to 3 providing a maximal score of 9, 21 and 9 for stress urinary incontinence, urge urinary incontinence and dysuria respectively. Women diagnosed with both stress and urge urinary incontinence by the USP were classified as having mixed urinary incontinence.
Prevalence of anal incontinence | 1 month
  The participant will be asked to fill out the anal incontinence Jorge and Wexner which contains five questions scored on a scale from zero (normal continence) to 20 (total incontinence).

SECONDARY OUTCOMES:
Risk factors for urinary and anal incontinence | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medecine, Monastir, Tunisia